CLINICAL TRIAL: NCT04658420
Title: A Single Ketamine Infusion Combined With Music for Suicidal Ideation During a Depressive Episode: A Randomized Open Label Clinical Trial
Brief Title: A Single Ketamine Infusion Combined With Music for Suicidal Ideation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Texas Health Science Center at Tyler (Other)
Collaborators: National Institutes of Health (NIH) (NIH); The University of Texas Health Science Center, Houston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2020-042; KL2TR003168 (NIH)
Record Dates: First submitted 2020-11-16; First posted 2020-12-08 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Suicidal Ideation; Depressive Episode
MeSH Terms: conditions — Suicidal Ideation | interventions — Ketamine; Music Therapy

STUDY DESIGN:
Intervention Model Description: All four groups will receive treatment as usual as defined above (potential approved hospitalization, medication, psychotherapy, outpatient referrals, suicide safety planning). A factorial design is being implemented to test four interventions. One group will receive IV ketamine 0.5mg/kg infused over forty minutes with one hour of pre-planned music will be compared to 3 other groups: One group will receive the same dose of ketamine without music, one group will one hour of music without ketamine, and one group will receive neither music nor ketamine. During the 4-week follow up interval, subjects from both groups will be contacted by phone for weekly assessment of depression, SI and quality of life.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Ketamine (Experimental): One group will receive IV ketamine 0.5mg/kg infused over forty minutes
  Interventions: Drug: Ketamine Hydrochloride
- Ketamine + Music (Experimental): One group will receive IV ketamine 0.5mg/kg infused over forty minutes with one hour of pre-planned music
  Interventions: Drug: Ketamine Hydrochloride; Other: Music
- Music (Experimental): One hour of pre-planned music without ketamine
  Interventions: Other: Music
- Treatment as usual (No Intervention): No music nor ketamine given

INTERVENTIONS:
Drug: Ketamine Hydrochloride — Individuals in the ketamine group will receive ketamine 0.5 mg/kg infused over 40 minutes
  Other Names: Ketamine
  Arms: Ketamine; Ketamine + Music
Other: Music — A playlist by composer Nils Frahm will be played for 60 minutes. The music is instrumental, relaxing and subjectively thought to be uplifting by patients who have listened to the music during ketamine infusions performed previously by the PI for treatment of resistant depression. Music can be previewed at the link below:
  https://open.spotify.com/playlist/37i9dQZF1DWVbGPBkXJYHF
  Arms: Ketamine + Music; Music

SUMMARY:
Suicidal ideation (SI) associated with major and bipolar depression is commonly seen in a wide range of clinical practice situations including the emergency room (ER). Current treatment regimens are often unsatisfactory. About a third of patients fail to respond to currently available therapy, and there are no currently FDA indicated rapid acting treatments for SI. Suboptimal outcomes have triggered the search for new, well-tolerated and more effective forms of treatment. Small clinical trials suggest that low dose (0.5mg/kg) ketamine is safe and effective for SI. We believe adding music during ketamine infusion may reduce anxiety and lead to more reduced SI based on available evidence. We are testing the hypothesis that a single infusion of ketamine combined with music enhances tolerability and improves outcomes in the treatment of SI when combined with treatment as usual in a factorial study design. One treatment with Ketamine + music will be compared to compared to one-time treatment with ketamine alone, music alone, or treatment as usual. 50 individuals with a depressive episode and suicidal ideation will receive intravenous (IV) ketamine 0.5mg/kg infused over 40 minutes once with 60 minutes of music, 50 individuals will receive IV ketamine without music, 50 subjects will receive 60 minutes of music once, and 50 patients will receive treatment as usual without ketamine or music. We anticipate that the ketamine + music group will have statistically significant indices of improvement in the primary outcome, suicidal ideation scores on the Scale for Suicidal Ideation (SSI) 4 weeks after the ketamine infusion. Secondary outcomes will include depression scores on the MontgomeryÅsberg Depression Rating Scale (MADRS) scale, adverse effects, and SSI scores at the end of 4 weeks. If, as we anticipate, the results indicate success of ketamine + music for SI, the work will identify new opportunities to more effectively manage patients with depression and suicidal ideation presenting to the ER.

DETAILED DESCRIPTION:
Ketamine is a glutamate N-methyl-D-aspartate (NMDA) receptor antagonist traditionally used as a general anesthetic. Recent double blinded randomized control trials of intravenous (IV) ketamine infusions have been well-tolerated and demonstrated a rapid onset of antidepressant effect, most notably in subjects with treatment-resistant depression (TRD) and treatment-resistant bipolar depression.

Significance. The outcomes of current therapy for depression are poor, with roughly a third of patient's failing to improve or regressing. The patients are high risk for suicide and the need for rapid acting, durable treatments for reduction of suicidal ideation is paramount.

Ketamine has been shown to improve suicidal ideation for at least 6 weeks in the largest study of ketamine for SI to date in subjects recruited to participate in the clinical trial and admitted to a research facility. We intend to test ketamine in a more pragmatic trial in the ER in patients who are not actively recruited, but report SI to ER staff or have SI as a chief complaint.

Research Aims.

Overview. In the current open label randomized control trial, we will examine the suicidal ideation reducing efficacy of IV ketamine combined with music and treatment as usual in four groups. All four groups will receive treatment as usual as defined above (potential hospitalization, medication, psychotherapy, outpatient referrals, suicide safety planning). A factorial design is being implemented to test two interventions independently and combined: ketamine and music. One group will receive IV ketamine 0.5mg/kg infused over forty minutes with one hour of pre-planned music will be compared to 3 other groups: One group will receive the same dose of ketamine without music, one group will one hour of music without ketamine, and one group will receive neither music nor ketamine. During the 4-week follow up interval, subjects from both groups will be contacted by phone for weekly assessment of depression, SI and quality of life.

A playlist by composer Nils Frahm will be played for 60 minutes. The music is instrumental, relaxing and subjectively thought to be uplifting by patients who have listened to the music during ketamine infusions performed previously by the PI for treatment of resistant depression. Music can be previewed at the link below:

https://open.spotify.com/playlist/37i9dQZF1DWVbGPBkXJYHF

Patients will be screened for study entry by the emergency room (ER) treating physician who will be available 24 hours a day who will notify the clinical trials research staff that a subject is available to be screened. Dr. Robert Creath Er attending will be the primary coordinator of Er services. The clinical trials staff that will be assigned to the project by the UTHET north campus department of clinical research. will then screen the subject for entry to the study, and perform the informed consent process. The subject will then be randomized by clinical trials staff using block randomization to each group. A 1:1 assignment to each group will be implemented with permuted blocks between 4 and 6 with equal probability. Patients entering the study will be voluntarily admitted to the hospital or monitored in the ER for a minimum of 2 hours after the first IV ketamine or music treatment and discharged when deemed to not be a suicide risk by a treating physician. A driver will be required to take the subject home if discharged the same day as the ketamine treatment. Subjects deemed to be a continued risk to themselves or others will be admitted as per clinician discretion which is considered treatment as usual. The ER nurse will be administering the sub-anesthetic dose of ketamine. Vital signs including, blood pressure, pulse oxygenation will be monitored at fifteen-minute intervals during the infusion, and will be recorded for 30 minutes after the infusion at fifteen minute intervals. Subjects will be followed up by phone at weekly intervals and voluntary hospitalization will be recommended for patients with SSI score of ≥4. Psychotropic medications will be adjusted and optimized at the discretion of the treating physicians at study entry. Medications may be modified during the 4-week study interval in line with standard practice. Informed consent will be obtained for all participants. Informed consent will be obtained in person when possible or by the Teams telemedicine app when necessary if research staff is unavailable on site.

The primary outcome measure of this study will be treatment response, defined as a ≥50% score reduction in the SSI from baseline to 4 weeks after the first ketamine injection. Remission will be defined as a ≥50% reduction in SSI score with score ≤4. The SSI will be administered at baseline, prior to each treatment and 24 hours after IV ketamine administration, then every week during the symptom monitoring follow-up period of 4 weeks. The clinician-rated SSI assesses current severity of suicidal ideation with 19 items scaled from 0 (least severe) to 2 (most severe). Medications may be adjusted during the study interval. Secondary outcome will be change in MADRS and SSI score from baseline to 4 weeks after the treatment. Raters will be blinded to the subject treatment group.

During the 4-week follow up participants will be contacted by phone with follow-up questions regarding their overall health status, mood and clinical state using MADRS, SSI, QIDS and other clinical scales listed below.

Study/Design. Patients with clinically documented depression with SI will be screened for diagnosis of depressive episode with the Mini-International Neuropsychiatric Interview (MINI), a structured interview of psychiatric disorders, at baseline to establish the presence of a major depressive episode. The depressive episode could be associated with major depressive disorder, bipolar disorder or substance induced depressive disorder.

Procedure

Portable speakers will be provided playing relaxing music prior to and during the administration of ketamine for groups 2 and 3 (Nils Frahm playlist-modern classical composer). This music has been previously used at Christus Mother Francis for therapeutic ketamine use with good results. Subjects will be inform that music can be stopped by request at any time. Informed consent and screening will be performed in the UTHET north campus clinical trials staff at initial presentation. Follow up assessments during weeks 1-4 will be done by phone. Clinical research staff will randomize subjects to treatment groups as documented above. Ketamine IV will be supplied by the UT Health East Texas pharmacy. The administration of ketamine will be initiated by the emergency room nurse with ACLS certified physician supervision.

Prior to the treatment, patients will be undergo psychiatric interview by the University of Texas Health center at Tyler psychiatric ER consult liaison team as per standard practice. An ACLS certified physician will be nearby in the ER post-procedure for 1 hour or until a clinician deems patient is clinically stable.

We plan on utilizing the monitoring protocol advised by the American Psychiatric Association consensus statement:

"(1) assessment of respiratory status (i.e., oxygen saturation or end-tidal CO2); (2) assessment of cardiovascular function (blood pressure and heart rate, reported on a regular basis every 15 minutes); (3) assessment of the level of consciousness or other documented assessment of responsiveness; and (4) delineation of criteria for stopping the infusion and a clear plan for managing cardiovascular or behavioral events during treatment."

Adverse events will be monitored and recorded throughout the study. The most common side effects associated with ketamine are nausea, vomiting, dizziness, double vision, drowsiness, elevated blood pressure, tachycardia, anxiety, dissociation (feeling strange and disconnected from the world), and confusion. Delirium, hallucinations, and nightmares have been associated with high dose ketamine, but are not common side effects in subanesthetic ketamine treatment. The subanesthetic dose of 0.5 mg/kg has been documented to be safe and well tolerated in numerous clinical trials in the treatment of suicidal thoughts.

Rare but serious possible adverse event associated with ketamine include:

Cardiac arrest, diabetes insipidus, anaphylaxis, ocular hypertension, increased intracranial pressure, arrythmia exacerbation or apnea.

Digital pulse oximetry, blood pressure, heart rate, and respiratory rate will be monitored throughout the injection at 15 minute intervals with a recovery period similar to recent study of IV ketamine for PTSD and TRD performed at the Minneapolis VA. Vital signs, the Clinician Administered Dissociative States Scale (CADSS) will be assessed pre-dose, at 40 minutes after ketamine infusion has started. Hypertensive emergency, respiratory failure or cardiac arrest is not known to have occurred in previous clinical trials of IV ketamine for treatment of depression. Emergency room physicians will be notified and render care in the event of unexpected medical emergencies. The infusions will be stopped if a patient requests stopping the infusion, becomes agitated, or goes into respiratory failure or cardiac arrest. Medical emergencies will be managed by ACLS certified ER physicians. Code BERT will be called as necessary if a patient becomes acutely agitated and presents a danger to themselves or others.

Medications will be optimized as per standard practice throughout the 4-week study. Suicide safety plans, referrals to outpatient treatments will done as per standard practice. Participants will be directed to contact the nearest ER in case of emergency after initial hospital discharge. Participants will be contacted weekly during the 4-week study period to review the patient's health status and administer clinical scales by phone.

Clinical assessment. Informed consent will be obtained. This evaluation will obtain family history and demographic data. We will perform a urine drug screening (UDS) to rule out recent undisclosed use of illicit substances that may exclude subjects from the study. Demographic information is obtained through a standardized form and covers age, race, gender, education (information both on siblings and their parents), religion, and socioeconomic status.

Participants will fill out the mood questionnaires rating the severity of the clinical symptoms. Participants will be asked about previous medications they have taken for mental health disorders and general medical conditions. Results will be stored in a secure location by the department of clinical research. Selected mood assessment questionnaires will be administered by our clinical research staff including the MINI Interview. This is the standard psychiatric research evaluation for ascertainment of psychiatric diagnosis in the context of research studies. It is a comprehensive structured interview for determining axis I diagnosis according to the DSM-V to be administered at study entry and takes approximately 15 minutes. We will also use the Montgomery Åsberg Depression Rating Scale (MADRS): this scale rates depressive symptoms, and its psychometric properties are well-established. We will assess SI with the Suicidal Scale Instrument. The clinician-rated SSI assessed current severity of suicidal ideation with 19 items scaled from 0 (least severe) to 2 (most severe). We will also assess dissociation with the Clinician-Administered Dissociative States Scale (CADSS): Frequency of administration: After every treatment, to monitor the dissociative side effects status post infusion.

Self-report questionnaires to assess mood, and quality of life will include Quick inventory of depressive symptomatology QIDS-SR to measure self-reported depressive symptoms, weekly and the World health organization quality of life scale.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18-64
* DSM-IV diagnosis of depressive episode as determined by the Mini International neuropsychiatric Interview criteria, and Montgomery Asberg Depression Rating Scale ≥ 28
* Suicidal ideation at baseline as and positive suicidal ideation defined as Scale for Suicidal Ideation score ≥4.
* Diagnosis of Major depressive disorder, bipolar disorder, or substance induced mood disorder will be included.

Exclusion Criteria:

* Active psychotic symptoms
* Current manic episode
* Previous diagnosis of Schizophrenia or Schizoaffective disorder
* Previous diagnosis of Intellectual disability or Autism Spectrum Disorder
* Previous diagnosis of Major Neurocognitive Disorder
* History of ketamine abuse or dependence
* Hypersensitivity to esketamine, ketamine, or any of the excipients.

Uncontrolled clinically significant medical conditions such as:

* Respiratory illness requiring the use of oxygen
* Previously documented prolonged QTc interval
* Current Aneurysmal vascular disease
* Arteriovenous malformation
* Intracerebral hemorrhage
* Unstable cardiac disease including history of myocardial infarction
* Positive urine pregnancy test
* Previous treatment of depression with Ketamine or Esketamine

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Scale for Suicide Ideation (SSI) | 4 weeks
  Clinician administered scale. Score range 0-38. Higher scores are indicative of increased suicidal ideation. The primary efficacy evaluation for each panel will be the change in SSI total score from baseline, prior to the first IV ketamine dose, to 4 weeks after IV ketamine treatment. 25 % reduction in score will be deemed treatment response, 50% reduction will be determined to be treatment remission.

SECONDARY OUTCOMES:
Montgomery Asberg Depression Rating Scale (MADRS) | 4 weeks
  Clinician administered depression rating scale. Score range= 0-60, higher scores are indicative of more severe depression. 50% score reduction is defined as response, 25% or less improvement in MADRS will be considered a non response.
World Health Organization Quality of life Scale (WHOQOL-BREF) | 4 weeks
  Score range- 0-100. Quality of life at study entry and every week. Higher scores are indicative of higher quality of life
Quick Inventory of Depressive Symptomatology (QIDS SR-16) | 4 weeks
  Self report measure of depression. Range 1-27, with higher scores indicative of more severe depression
Time of hospitalization | 4 weeks
  Average days of hospitalization between treatment groups

CONTACTS AND LOCATIONS:
Overall Officials: Richard Idell, MD, Principal Investigator — University of Texas Health Science Center at Tyler
Locations (1):
- UT Health East Texas, Tyler, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fava M. Diagnosis and definition of treatment-resistant depression. Biol Psychiatry. 2003 Apr 15;53(8):649-59. doi: 10.1016/s0006-3223(03)00231-2. PMID 12706951
- [Background] Rush AJ, Trivedi MH, Wisniewski SR, Nierenberg AA, Stewart JW, Warden D, Niederehe G, Thase ME, Lavori PW, Lebowitz BD, McGrath PJ, Rosenbaum JF, Sackeim HA, Kupfer DJ, Luther J, Fava M. Acute and longer-term outcomes in depressed outpatients requiring one or several treatment steps: a STAR*D report. Am J Psychiatry. 2006 Nov;163(11):1905-17. doi: 10.1176/ajp.2006.163.11.1905. PMID 17074942
- [Background] Grunebaum MF, Ellis SP, Keilp JG, Moitra VK, Cooper TB, Marver JE, Burke AK, Milak MS, Sublette ME, Oquendo MA, Mann JJ. Ketamine versus midazolam in bipolar depression with suicidal thoughts: A pilot midazolam-controlled randomized clinical trial. Bipolar Disord. 2017 May;19(3):176-183. doi: 10.1111/bdi.12487. Epub 2017 Apr 28. PMID 28452409
- [Background] aan het Rot M, Collins KA, Murrough JW, Perez AM, Reich DL, Charney DS, Mathew SJ. Safety and efficacy of repeated-dose intravenous ketamine for treatment-resistant depression. Biol Psychiatry. 2010 Jan 15;67(2):139-45. doi: 10.1016/j.biopsych.2009.08.038. PMID 19897179
- [Background] Wilkinson ST, Ballard ED, Bloch MH, Mathew SJ, Murrough JW, Feder A, Sos P, Wang G, Zarate CA Jr, Sanacora G. The Effect of a Single Dose of Intravenous Ketamine on Suicidal Ideation: A Systematic Review and Individual Participant Data Meta-Analysis. Am J Psychiatry. 2018 Feb 1;175(2):150-158. doi: 10.1176/appi.ajp.2017.17040472. Epub 2017 Oct 3. PMID 28969441
- [Background] Grunebaum MF, Galfalvy HC, Choo TH, Keilp JG, Moitra VK, Parris MS, Marver JE, Burke AK, Milak MS, Sublette ME, Oquendo MA, Mann JJ. Ketamine for Rapid Reduction of Suicidal Thoughts in Major Depression: A Midazolam-Controlled Randomized Clinical Trial. Am J Psychiatry. 2018 Apr 1;175(4):327-335. doi: 10.1176/appi.ajp.2017.17060647. Epub 2017 Dec 5. PMID 29202655
- [Background] George D, Galvez V, Martin D, Kumar D, Leyden J, Hadzi-Pavlovic D, Harper S, Brodaty H, Glue P, Taylor R, Mitchell PB, Loo CK. Pilot Randomized Controlled Trial of Titrated Subcutaneous Ketamine in Older Patients with Treatment-Resistant Depression. Am J Geriatr Psychiatry. 2017 Nov;25(11):1199-1209. doi: 10.1016/j.jagp.2017.06.007. Epub 2017 Jun 13. PMID 28739263
- [Background] Aalbers S, Fusar-Poli L, Freeman RE, Spreen M, Ket JC, Vink AC, Maratos A, Crawford M, Chen XJ, Gold C. Music therapy for depression. Cochrane Database Syst Rev. 2017 Nov 16;11(11):CD004517. doi: 10.1002/14651858.CD004517.pub3. PMID 29144545
- [Background] Bradt J, Dileo C, Shim M. Music interventions for preoperative anxiety. Cochrane Database Syst Rev. 2013 Jun 6;2013(6):CD006908. doi: 10.1002/14651858.CD006908.pub2. PMID 23740695
- [Background] Feder A, Parides MK, Murrough JW, Perez AM, Morgan JE, Saxena S, Kirkwood K, Aan Het Rot M, Lapidus KA, Wan LB, Iosifescu D, Charney DS. Efficacy of intravenous ketamine for treatment of chronic posttraumatic stress disorder: a randomized clinical trial. JAMA Psychiatry. 2014 Jun;71(6):681-8. doi: 10.1001/jamapsychiatry.2014.62. PMID 24740528
- [Background] Mithoefer MC, Mithoefer AT, Feduccia AA, Jerome L, Wagner M, Wymer J, Holland J, Hamilton S, Yazar-Klosinski B, Emerson A, Doblin R. 3,4-methylenedioxymethamphetamine (MDMA)-assisted psychotherapy for post-traumatic stress disorder in military veterans, firefighters, and police officers: a randomised, double-blind, dose-response, phase 2 clinical trial. Lancet Psychiatry. 2018 Jun;5(6):486-497. doi: 10.1016/S2215-0366(18)30135-4. Epub 2018 May 1. PMID 29728331
- [Background] Carhart-Harris RL, Bolstridge M, Rucker J, Day CM, Erritzoe D, Kaelen M, Bloomfield M, Rickard JA, Forbes B, Feilding A, Taylor D, Pilling S, Curran VH, Nutt DJ. Psilocybin with psychological support for treatment-resistant depression: an open-label feasibility study. Lancet Psychiatry. 2016 Jul;3(7):619-27. doi: 10.1016/S2215-0366(16)30065-7. Epub 2016 May 17. PMID 27210031
- [Background] Albott CS, Lim KO, Forbes MK, Erbes C, Tye SJ, Grabowski JG, Thuras P, Batres-Y-Carr TM, Wels J, Shiroma PR. Efficacy, Safety, and Durability of Repeated Ketamine Infusions for Comorbid Posttraumatic Stress Disorder and Treatment-Resistant Depression. J Clin Psychiatry. 2018 May/Jun;79(3):17m11634. doi: 10.4088/JCP.17m11634. PMID 29727073
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Montgomery SA, Asberg M. A new depression scale designed to be sensitive to change. Br J Psychiatry. 1979 Apr;134:382-9. doi: 10.1192/bjp.134.4.382. PMID 444788
- [Background] Beck AT, Kovacs M, Weissman A. Assessment of suicidal intention: the Scale for Suicide Ideation. J Consult Clin Psychol. 1979 Apr;47(2):343-52. doi: 10.1037//0022-006x.47.2.343. No abstract available. PMID 469082
- See also: The Underlying Cause of Death database contains mortality and population counts for all U.S. counties. Data are based on death certificates for U.S. residents. — http://wonder.cdc.gov/ucd-icd10.html
- See also: Smith county Suicide rates — http://www.census.gov/quickfacts/smithcountytexas